CLINICAL TRIAL: NCT04976439
Title: Genomic Landscape of APC, KRAS, TP53, PIK3CA, and MLH1 in Colorectal
Brief Title: Patogenic Mutation in 5 Genes
Status: Completed | Type: Observational
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Vania Myralda Giamour Marbun, Principal Investigator - Staff of Digestive Division - General Surgery Department, Dr Cipto Mangunkusumo General Hospital
Other Study IDs: MUTASICRC
Record Dates: First submitted 2021-07-02; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Cancer; APC Gene Mutation; TP53 Gene Mutation; PIK3CA Gene Mutation; KRAS Mutation-Related Tumors; MLH1 Gene Mutation
Keywords: next-generation sequencing; colorectal cancer; indonesia population; co-occurring mutation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Age
  Interventions: Other: co-occuring mutation
- Grade
  Interventions: Other: co-occuring mutation
- Tumor location
  Interventions: Other: co-occuring mutation
- Stage
  Interventions: Other: co-occuring mutation
- Lymphovascular invasion
  Interventions: Other: co-occuring mutation

INTERVENTIONS:
Other: co-occuring mutation — APC, TP53, PIK3CA, KRAS APC, TP53, PIK3CA, MLH1 APC, TP53, PIK3CA, KRAS, and MLH1 APC, TP53, PIK3CA

SUMMARY:
This is a pathogenic mutation profile of colorectal patients specifically in 5 genes, i.e. APC, TP53, PIK3CA, KRAS, and MLH1. Single nucleotide variants identified were synchronized with patients' characteristics.

ELIGIBILITY:
Inclusion Criteria:

* FFPE samples fullfilling purity criterion and pass quality control

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a descriptive study in patients with colorectal malignancies who underwent surgery and/or chemoradiation and/or chemotherapy at RSCM, RSKJ, and MRCCC in 2017-2018 whose tumor tissue specimens were still properly stored in the form of formalin-fixed paraffin-embedded (FFPE). .
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Description of clinical characteristics | January 2017 - June 2021
  Age, gender
Description of tumor nature | January 2017 - June 2021
  grade, stage, lymphovascular invasion, tumor location
Description of survival | January 2017 - June 2021
  Median of life expectancy

CONTACTS AND LOCATIONS:
Locations (1):
- Vania Myralda Giamour Marbun, Jakarta, ALL, Indonesia

IPD SHARING:
Plan to Share IPD: No